CLINICAL TRIAL: NCT01849172
Title: Effect and Safety of Electroacupuncture for Symptoms of Menopausal Transition -a Multicenter Randomized Controlled Trial
Brief Title: Effect and Safety of Electroacupuncture for Symptoms of Menopausal Transition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Principal Investigator, Liu Zhishun, Dean of Acupuncture Department of Guangan'men Hospital, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BAI24B01
Record Dates: First submitted 2013-05-05; First posted 2013-05-08 (Estimated); Results first posted 2019-03-25 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Menopausal Syndrome
MeSH Terms: interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- electroacupuncture (Experimental): Electroacupuncture at RN4, EX-CA1，ST25, SP6 (double sides). One session will be given every two days, 3 sessions per week (24 sessions in all) and each session lasts for 30 minutes.
  Interventions: Other: electroacupuncture
- sham electroacupuncture (Sham Comparator): Sham electroacupuncture at non-points proximate to RN4 (P1), EX-CA1(P2)，ST25 (P3) and SP6 (P4) (double sides).Specially constructed EA apparatus were used with no skin penetration, electricity output, or de qi requirement for needle manipulation One session will be given every two days, 3 sessions per week (24 sessions in all) and each session lasts for 30 minutes.
  Interventions: Other: sham electroacupuncture

INTERVENTIONS:
Other: electroacupuncture — Stick adhesive tapes to all points. For ST25, EX-CA1 and RN4, insert the needle vertically through the pads and the skin, and then slowly and vertically penetrate through the layer of fatty tissue, into the muscles of the abdominal wall .For RN4, manipulate the needle with an even lifting, thrusting and twisting method slightly for 3 times. Insert the needle vertically at SP6 to a depth of 1 cm. Manipulate the needle with an even lifting, thrusting and twisting method slightly for 3 times to reach de-qi. Put the electric stimulator on the pair of EX-CA1 and ST25 points with a dilatational wave, 10/50 Hz, 0.5-1.0mA. To turn on the current intensity till the abdomen shivers. The same manipulation methods for RN4 and SP6 will be given every 10 minutes (3 times in all).
  Arms: electroacupuncture
Other: sham electroacupuncture — Non-points proximate to RN4 (P1), EX-CA1(P2)，ST25 (P3) and SP6 (P4) (double sides) are used.P1 and P3 are at the sites 1 cm (outward in horizontal direction) proximate to RN4 and ST25 respectively. P2 is 2 cm (outward in horizontal direction) proximate to EX-CA1. P4 is at the middle site of the spleen meridian and the kidney meridian (backward in horizontal direction proximate to SP6).
  Stick adhesive tapes to all points. Blunt needles will be used to be inserted to but not piercing the skin. Even lifting, thrusting and twisting manipulation methods will be given for each non-point for 3 times. Put the sham electric stimulator on the pair of P2 and P3 with the same parameters as the acupuncture group. But there is no current intensity actually.
  Arms: sham electroacupuncture

SUMMARY:
The primary object is to evaluate the efficacy and safety of electroacupuncture for symptoms of women during menopausal transition .

DETAILED DESCRIPTION:
Menopause transition is called perimenopause in the past time. 40-80% women aged 40 to 65 have symptoms during this period. Hormone therapy is the recommended therapy for menopause and there is not enough evidence in favor of alternative medicine's effect.

Our pilot trial showed that electroacupuncture had better effect for menopause transition symptoms than sham electroacupuncture. We are going to conduct a phase Ⅱ clinical trial to further evaluate the safety and effect of electroacupuncture for menopause transition symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Cycle irregularity (periods occur 7 days or over earlier or later ) in the past 12 months (early menopausal transition); subjects with the last menstruation at least 2 but no longer than 12 months in the past 12 months (late menopausal transition).
2. Menopausal transition symptoms such as hot flushes, sweating, sleep disturbance, migraine, anxiety, vaginal dryness and sexual problems.
3. 40 to 55 years old.
4. Volunteer to join in the trial and sign the informed consent. Patients conformed with the 4 items at the same time will be included. -

Exclusion Criteria:

1. Regular cycles during the past 3 months before enrollment.
2. use of estrogen, SSRIs, soybean isoflavone, progestin, vitamin E or black sesame in the past 4 weeks.
3. Patients with ovarian cyst, uterine myoma (diameter≥4cm) or after hysterectomy/ ovariectomy.
4. Patients with radiochemotherapy history or undergoing radiochemotherapy.
5. Cryptogenic vaginal bleeding
6. Coagulation disorder or use of anticoagulants like warfarin and heparin sodium.
7. Existing skin diseases like eczema or psoriasis.
8. Severe hepatic/renal insufficiency.
9. Insufficiently controlled hypertension, diabetes or thyroid diseases.
10. Existing diabetic neuropathy, malignant tumor and psychiatric disorders.
11. Wish to become pregnant or is pregnant or breast-feeding.
12. Regular use of sedative or anxiolytic.
13. Smoking or alcohol intake.
14. Subjects with mandatory indication for HT (e.g. postsurgical menopause or active osteoporosis).
15. With cardiac pacemaker or artificial joint.

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 360 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhishun Liu, Ph.D, Study Chair — Guang'an Men Hospital Affiliated to China Academy of Chinese Medical Sciences
Locations (1):
- Guangan'men Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu Z, Wang Y, Xu H, Wu J, He L, Jiang JY, Yan S, Du R, Liu B. Efficacy of electroacupuncture for symptoms of menopausal transition: study protocol for a randomized controlled trial. Trials. 2014 Jun 21;15:242. doi: 10.1186/1745-6215-15-242. PMID 24950841

RESULTS

PARTICIPANT FLOW:
Groups:
- Acupuncture: Electroacupuncture at RN4, EX-CA1，ST25, SP6 (double sides). One session will be given every two days, 3 sessions per week (24 sessions in all) and each session lasts for 30 minutes.
  acupuncture: Stick adhesive tapes to all points. For ST25, EX-CA1 and RN4, insert the needle vertically through the pads and the skin, and then slowly and vertically penetrate through the layer of fatty tissue, up into the muscles of the abdominal wall .For RN4, manipulate the needle with an even lifting, thrusting and twisting method slightly for 3 times. Insert the needle vertically at SP6 to a depth of 1 cm. Manipulate the needle with an even lifting, thrusting and twisting method slightly for 3 times to reach de-qi. Put the electric stimulator on the pair of EX-CA1 and ST25 points with a dilatational wave, 10/50 Hz, 0.5-1.0mA. To turn on the current intensity till the abdomen shivers. The same manipulation methods for RN4 and SP6 will be given every 10 minutes (3 times in all).
- Sham Acupuncture: Electroacupuncture at non-points proximate to RN4 (P1), EX-CA1(P2)，ST25 (P3) and SP6 (P4) (double sides).
  One session will be given every two days, 3 sessions per week (24 sessions in all) and each session lasts for 30 minutes.
  sham acupuncture: Non-points proximate to RN4 (P1), EX-CA1(P2)，ST25 (P3) and SP6 (P4) (double sides) are used.P1 and P3 are at the sites 1 cm (outward in horizontal direction) proximate to RN4 and ST25 respectively. P2 is 2 cm (outward in horizontal direction) proximate to EX-CA1. P4 is at the middle site of the spleen meridian and the kidney meridian (backward in horizontal direction proximate to SP6).
  Stick adhesive tapes to all points. Blunt needles will be used to be inserted to but not piercing the skin. Even lifting, thrusting and twisting manipulation methods will be given for each non-point for 3 times. Put the sham electric stimulator on the pair of P2 and P3 with the same parameters as the acupuncture group. But there is no current intensity actu
Period: Overall Study
Arm/Group | Acupuncture | Sham Acupuncture
Started | 180 | 180
Completed | 173 | 174
Not Completed | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Sham Acupuncture: Electroacupuncture at non-points proximate to RN4 (P1), EX-CA1(P2)，ST25 (P3) and SP6 (P4) (double sides).One session will be given every two days, 3 sessions per week (24 sessions in all) and each session lasts for 30 minutes.
  sham acupuncture: Non-points proximate to RN4 (P1), EX-CA1(P2)，ST25 (P3) and SP6 (P4) (double sides) are used.P1 and P3 are at the sites 1 cm (outward in horizontal direction) proximate to RN4 and ST25 respectively. P2 is 2 cm (outward in horizontal direction) proximate to EX-CA1. P4 is at the middle site of the spleen meridian and the kidney meridian (backward in horizontal direction proximate to SP6).Stick adhesive tapes to all points. Blunt needles will be used to be inserted to but not piercing the skin. Even lifting, thrusting and twisting manipulation methods will be given for each non-point for 3 times. Put the sham electric stimulator on the pair of P2 and P3 with the same parameters as the acupuncture group. But there is no current intensity actual
- Total: Total of all reporting groups
Arm/Group | Acupuncture | Sham Acupuncture | Total
Number analyzed (Participants) | 180 | 180 | 360
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 180 | 180 | 360
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 48.7 (4.0) | 48.1 (3.8) | 48.4 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 180 | 180 | 360
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 180 | 180 | 360

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Menopause Rating Scale Total Score
Description: The change in menopause rating scale (MRS) total score compared with baseline at week 8 equals MRS total score at week 8 minus MRS total score at baseline.
  MRS is a self-report questionnaire for evaluating the severity of menopausal symptoms in women, which contains 11 items. Each of the 11 symptoms contained a scoring scale from "0" (no complaints) to "4" (very severe symptoms). The total score will be calculated as the all items ranging from 0 to 44, with higher scores indicating worse symptoms. The MRS including 3 dimensions: psychological, somatic-vegetative, and urogenital.
Time Frame: at baseline and week 8
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Electroacupuncture: Acupoints of RN4, Bilateral EX-CA1, ST25 and SP 6 were used.For acupoints in the abdomen, the needles will be inserted vertically and then slowly and vertically penetrate through the layer of fatty tissue, up into the muscles of the abdominal wall. The needle will be inserted vertically at SP6 to a depth of 1 cun. Paired alligator clips of the EA apparatus will be attached transversely to the needle holders of the bilateral EX-CA1 and ST25. EA stimulation will last for 30 minutes with a dilatational wave of 10/50Hz and current intensity of 0.1 to 1mA. The current intensity will be increased until the skin around the acupoints shivers. The manipulation on RN4 and SP6 mentioned above should be performed every 10 minutes, three times in 30 minutes.Patients will be treated with EA 3 sessions a week on alternate days for 8 successive weeks, 24 sessions for each patient in total.
- Sham Electroacupuncture: Non-points proximate to RN4 , EX-CA1，ST25 and SP6 were used. After sterilizing the skin, placebo needles of size 0.30×25 mm will be needled into adhesive pads without skin penetration or needle manipulation. The needle will be manipulated slightly with an even lifting, thrusting, and twisting method repeated three times for each point but no deqi. Paired alligator clips of the specially made EA apparatus (power output lines, which connect the alligator clips and the EA apparatus, will be cut inside with an appearance as usual) will be attached transversely to the needle holders of the bilateral sham-ST25 and sham-EX-CA1. The EA apparatus will be turned on with a working power indicator and the same sound as the EA group. The parameters of sham EA apparatus and the treatment course will be the same as in the EA group.
Arm/Group | Electroacupuncture | Sham Electroacupuncture
Number analyzed (Participants) | 180 | 180
units on a scale | 6.3 [5.0 to 7.7] | 4.5 [3.2 to 5.8]
Statistical Analysis 1: Comparison: Electroacupuncture vs Sham Electroacupuncture; Test type: Superiority; p = 0.05, Mixed Models Analysis

2. Secondary Outcome: Change From Baseline in Menopause Rating Scale Total Score
Description: The change in Menopause Rating Scale (MRS）total score compared with baseline at weeks 4, 20 and 32 equals MRS total score at weeks 4, 20 and 32 minus MRS total score at baseline,respectively.
  MRS is a self-report questionnaire for evaluating the severity of menopausal symptoms in women, which contains 11 items. Each of the 11 symptoms contained a scoring scale from "0" (no complaints) to "4" (very severe symptoms). The total score will be calculated as the all items ranging from 0 to 44, with higher scores indicating worse symptoms. The MRS including 3 dimensions: psychological, somatic-vegetative, and urogenital.
Time Frame: at baseline，and weeks 4, 20 and 32
Population: 6 participants in the electroacupuncture group and 5 participants in the sham electroacupuncture group were missing at week 4 and week 8.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Electroacupuncture | Sham Electroacupuncture
Number analyzed (Participants) | 174 | 175
units on a scale
  Change at week 4 | 3.6 [2.6 to 4.6] | 3.2 [2.2 to 4.2]
  Change at week 20: number analyzed (Participants) | 173 | 174
  Change at week 20 | 7.0 [5.5 to 8.4] | 4.5 [3.1 to 5.9]
  Change at week 32: number analyzed (Participants) | 173 | 174
  Change at week 32 | 6.8 [5.2 to 8.5] | 4.1 [2.5 to 5.8]

3. Secondary Outcome: Change From Baseline in Somatic-vegetative Domain of Menopause Rating Scale
Description: The change from baseline in somatic-vegetative domain of Menopause Rating Scale(MRS) at weeks 4, 8, 20 and 32 equals the somatic-vegetative domain of MRS at weeks 4, 8, 20 and 32 minus the somatic-vegetative domain of MRS at baseline, respectively.
  The somatic-vegetative domain contains 4 items (items 1-3 and 11). Each of the item scores ranges from 0 to 4. The somatic-vegetative domain score will be calculated as the all somatic-vegetative items ranging from 0 to 16, with higher scores indicating worse symptoms.
Time Frame: at baseline, and weeks 4, 8, 20 and 32
Population: 6 participants in the electroacupuncture group and 5 participants in the sham electroacupuncture group were missing at week 4 and week 8. 7 participants in the electroacupuncture group and 6 participants in the sham electroacupuncture group were missing at week 20 and week 32
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Electroacupuncture | Sham Electroacupuncture
Number analyzed (Participants) | 174 | 175
units on a scale
  Change at week 4 | 1.5 [1.1 to 2.0] | 1.4 [1.0 to 1.8]
  Change at week 8 | 2.6 [2.0 to 3.2] | 1.9 [1.4 to 2.5]
  Change at week 20: number analyzed (Participants) | 173 | 174
  Change at week 20 | 3.0 [2.4 to 3.5] | 2.0 [1.5 to 2.5]
  Change at week 32: number analyzed (Participants) | 173 | 174
  Change at week 32 | 2.8 [2.2 to 3.4] | 1.7 [1.2 to 2.3]

4. Secondary Outcome: Change From Baseline in Psychological Domain of Menopause Rating Scale
Description: The change from baseline in psychological domain of Menopause Rating Scale(MRS) at weeks 4, 8, 20 and 32 equals the psychological domain of MRS at weeks 4, 8, 20 and 32 minus the psychological domain of MRS at baseline, respectively.
  The psychological domain contains 4 items (items 4-7). Each of the item scores ranges from 0 to 4. The psychological domain score will be calculated as the all psychological items ranging from 0 to 16, with higher scores indicating worse symptoms.
Time Frame: at baseline, and weeks 4, 8, 20 and 32
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Electroacupuncture | Sham Electroacupuncture
Number analyzed (Participants) | 174 | 175
units on a scale
  Change at week 4 | 1.6 [1.1 to 2.1] | 1.5 [1.0 to 2.0]
  change at week 8 | 2.7 [2.1 to 3.3] | 2.0 [1.4 to 2.6]
  change at week 20: number analyzed (Participants) | 173 | 174
  change at week 20 | 2.9 [2.2 to 3.6] | 2.0 [1.3 to 2.7]
  Change at week 32: number analyzed (Participants) | 173 | 174
  Change at week 32 | 3.0 [2.2 to 3.7] | 2.0 [1.3 to 2.8]

5. Secondary Outcome: Change From Baseline in Urogenital Domain of Menopause Rating Scale
Description: The change from baseline in urogenital domain of Menopause Rating Scale(MRS) at weeks 4, 8, 20 and 32 equals the urogenital domain of MRS at weeks 4, 8, 20 and 32 minus the urogenital domain of MRS at baseline, respectively.
  The urogenital domain contains 3 items (items 8-10). Each of the item scores ranges from 0 to 4. The psychological domain score will be calculated as the all urogenital items ranging from 0 to 12, with higher scores indicating worse symptoms.
Time Frame: at baseline, and weeks 4, 8, 20 and 32
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Electroacupuncture | Sham Electroacupuncture
Number analyzed (Participants) | 174 | 175
units on a scale
  Change at week 4 | 0.5 [0.2 to 0.7] | 0.3 [0.1 to 0.6]
  Change at week 8 | 1.0 [0.7 to 1.4] | 0.5 [0.2 to 0.8]
  Change at week 20: number analyzed (Participants) | 173 | 174
  Change at week 20 | 1.1 [0.7 to 1.5] | 0.5 [0.1 to 0.9]
  Change at week 32: number analyzed (Participants) | 173 | 174
  Change at week 32 | 1.0 [0.6 to 1.5] | 0.4 [-0.1 to 0.9]

6. Secondary Outcome: Change From Baseline in Mean 24-h Hot Flash Score
Description: The 24-h hot flash score was daily hot flash episodes multiplied by the corresponding severities. The change from baseline in mean 24-h HF score at weeks 4, 8, 20 and 32 equals the mean 24-h HF score at weeks 4 , 8, 20 and 32 minus the mean 24-h HF score at baseline, respectively.
  Hot flashes score consisted the number and the degree of hot flashes. The hot flashes score is the sum of the scores of all the hot flashes occurring in a whole day, with a higher score indicating worse symptoms. A 3-point rating scale allows the women to describe the perceived severity of hot flash. 1 point = mild hot flash, 2 point = moderate hot flash, 3 point = severe hot flash.
Time Frame: at baseline, and weeks 4, 8, 20 and 32
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Electroacupuncture | Sham Electroacupuncture
Number analyzed (Participants) | 174 | 175
units on a scale
  Change at week 4 | 1.9 [1.0 to 2.8] | 1.9 [0.9 to 2.8]
  Change at week 8 | 3.6 [2.6 to 4.7] | 2.5 [1.4 to 3.5]
  Change at week 20: number analyzed (Participants) | 173 | 174
  Change at week 20 | 3.9 [2.9 to 4.8] | 2.7 [1.7 to 3.7]
  Change at week 32: number analyzed (Participants) | 173 | 174
  Change at week 32 | 4.1 [2.7 to 5.5] | 1.9 [0.5 to 3.2]

7. Secondary Outcome: Change From Baseline in Menopause-Specific Quality of Life Questionnaire Total Score
Description: The change from baseline in Menopause-Specific Quality of Life Questionnaire (MENQOL) total score at weeks 4, 8, 20 and 32 equals the MENQOL total score at weeks 4, 8, 20 and 32 minus the MENQOL score at baseline, respectively.
  It composed of 29 items and was divided into four domains: vasomotor (items 1-3), psychosocial (items 4-10), physical (items 11-26), and sexual (items 27-29). Each of the item scores ranges from 0 to 6. The total score will be calculated as the all items ranging from 0 to 174, with lower scores indicating a better quality of life.
Time Frame: at baseline, and weeks 4, 8, 20 and 32
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Electroacupuncture | Sham Electroacupuncture
Number analyzed (Participants) | 174 | 175
units on a scale
  Change at week 4 | 12.8 [8.6 to 17.0] | 12.6 [8.4 to 16.8]
  Change at week 8 | 22.8 [16.9 to 28.7] | 17.1 [11.2 to 23]
  Change at week 20: number analyzed (Participants) | 173 | 174
  Change at week 20 | 25.3 [18.9 to 31.7] | 18.2 [11.9 to 24.6]
  Change at week 32: number analyzed (Participants) | 173 | 174
  Change at week 32 | 26 [19.4 to 32.7] | 17.6 [11.0 to 24.3]

8. Secondary Outcome: Change From Baseline in the Vasomotor Domain of Menopause-Specific Quality of Life Questionnaire
Description: The change from baseline in the vasomotor domain of Menopause-Specific Quality of Life Questionnaire (MENQOL) at weeks 4, 8, 20 and 32 equals the vasomotor domain of MENQOL at weeks 4, 8, 20 and 32 minus the vasomotor domain of MENQOL at baseline, respectively.
  The vasomotor domain contains 3 items (items 1-3). Each of the item scores ranges from 0 to 6. The vasomotor domain score will be calculated as the all vasomotor items ranging from 0 to 18, with lower scores indicating a better quality of life.
Time Frame: at baseline, and weeks 4, 8, 20 and 32
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Electroacupuncture | Sham Electroacupuncture
Number analyzed (Participants) | 174 | 175
units on a scale
  Change at week 4 | 1.9 [1.1 to 2.8] | 1.7 [0.9 to 2.6]
  Change at week 8 | 3.4 [2.4 to 4.4] | 2.5 [1.5 to 3.5]
  Change at week 20: number analyzed (Participants) | 173 | 174
  Change at week 20 | 3.7 [2.7 to 4.7] | 2.7 [1.6 to 3.7]
  Change at week 32: number analyzed (Participants) | 173 | 174
  Change at week 32 | 3.8 [2.8 to 4.8] | 2.4 [1.4 to 3.4]

9. Secondary Outcome: Change From Baseline in the Psychosocial Domain of Menopause-Specific Quality of Life Questionnaire
Description: The change from baseline in the psychosocial domain of Menopause-Specific Quality of Life Questionnaire (MENQOL) at weeks 4, 8, 20 and 32 equals the psychosocial domain of MENQOL at weeks 4, 8, 20 and 32 minus the psychosocial domain of MENQOL at baseline, respectively.
  The psychosocial domain contains 7 items (items 4-10). Each of the item scores ranges from 0 to 6. The vasomotor domain score will be calculated as the all psychosocial items ranging from 0 to 42, with lower scores indicating a better quality of life.
Time Frame: at baseline, and weeks 4, 8, 20 and 32
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Electroacupuncture | Sham Electroacupuncture
Number analyzed (Participants) | 174 | 175
units on a scale
  Change at week 4 | 2.8 [1.7 to 4.0] | 2.8 [1.7 to 4.0]
  Change at week 8 | 5.5 [4.0 to 7.0] | 3.8 [2.4 to 5.3]
  Change at week 20: number analyzed (Participants) | 173 | 174
  Change at week 20 | 6.1 [4.4 to 7.9] | 4.2 [2.5 to 6.0]
  Change at week 32: number analyzed (Participants) | 173 | 174
  Change at week 32 | 6.4 [4.5 to 8.3] | 4.3 [2.4 to 6.2]

10. Secondary Outcome: Change From Baseline in the Physical Domain of Menopause-Specific Quality of Life Questionnaire
Description: The change from baseline in the physical domain of Menopause-Specific Quality of Life Questionnaire (MENQOL) at weeks 4, 8, 20 and 32 equals the physical domain of MENQOL at weeks 4, 8, 20 and 32 minus the physical domain of MENQOL at baseline, respectively.
  The physical domain contains 16 items (items 11-26). Each of the item scores ranges from 0 to 6. The vasomotor domain score will be calculated as the all physical items ranging from 0 to 96, with lower scores indicating a better quality of life.
Time Frame: at baseline, and weeks 4, 8, 20 and 32
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Electroacupuncture | Sham Electroacupuncture
Number analyzed (Participants) | 174 | 175
units on a scale
  Change at week 4 | 7.4 [4.7 to 9.6] | 7.3 [4.9 to 9.7]
  Change at week 8 | 12.4 [9.1 to 15.8] | 9.5 [6.2 to 12.9]
  Change at week 20: number analyzed (Participants) | 173 | 174
  Change at week 20 | 14.1 [10.6 to 17.6] | 10.1 [6.6 to 13.7]
  Change at week 32: number analyzed (Participants) | 173 | 174
  Change at week 32 | 14.3 [10.7 to 18.0] | 10.0 [6.4 to 13.6]

11. Secondary Outcome: Change From Baseline in the Sexual Functioning Domain of Menopause-Specific Quality of Life Questionnaire
Description: The change from baseline in the sexual functioning domain of Menopause-Specific Quality of Life Questionnaire (MENQOL) at weeks 4, 8, 20 and 32 equals the sexual functioning domain of MENQOL at weeks 4, 8, 20 and 32 minus the sexual functioning domain of MENQOL at baseline, respectively.
  The sexual functioning domain contains 3 items (items 27-29). Each of the item scores ranges from 0 to 6. The vasomotor domain score will be calculated as the all sexual functioning items ranging from 0 to 18, with lower scores indicating a better quality of life.
Time Frame: at baseline, and weeks 4, 8, 20 and 32
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Electroacupuncture | Sham Electroacupuncture
Number analyzed (Participants) | 174 | 175
units on a scale
  Change at week 4 | 0.9 [0.5 to 1.3] | 0.8 [0.4 to 1.2]
  Change at week 8 | 1.5 [1.0 to 1.9] | 1.2 [0.7 to 1.6]
  Change at week 20: number analyzed (Participants) | 173 | 174
  Change at week 20 | 1.4 [0.8 to 1.9] | 1.2 [0.6 to 1.7]
  Change at week 32: number analyzed (Participants) | 173 | 174
  Change at week 32 | 1.5 [0.7 to 2.2] | 1.0 [0.2 to 1.8]

12. Secondary Outcome: Change From Baseline in Serum FSH Level
Description: The change from baseline in serum FSH level at weeks 8 and 20 equals FSH at weeks 8 and 20 minus FSH at baseline, respectively.
Time Frame: at baseline, and weeks 8 and 20
Population: FSH, LH, and FSH/LH values were missing in 9 participants in the electroacupuncture group and 8 participants in the sham electroacupuncture group at week 8, and in 16 participants in the electroacupuncture group and 14 participants in the sham electroacupuncture group at week 20.
Measure: Mean (95% Confidence Interval); unit: mIU/ml
Arm/Group | Electroacupuncture | Sham Electroacupuncture
Number analyzed (Participants) | 171 | 172
mIU/ml
  Change at week 8 | 4.1 [0.4 to 7.9] | 2.0 [-1.8 to 5.9]
  Change at week 20: number analyzed (Participants) | 164 | 166
  Change at week 20 | 0.6 [-0.4 to 5.3] | 0.4 [-3.7 to 4.6]

13. Secondary Outcome: Change From Baseline in Serum E2 Level
Description: The change from baseline in serum E2 level at weeks 8 and 20 equals E2 at weeks 8 and 20 minus E2 at baseline, respectively.
Time Frame: at baseline, and weeks 8 and 20
Population: Estradiol values were missing in 37 participants in the electroacupuncture group and 39 participants in the sham electroacupuncture group at week 8, and in 44 patients in the electroacupuncture group and 38 participants in the sham electroacupuncture group at week 20.
Measure: Mean (95% Confidence Interval); unit: pmol/ml
Arm/Group | Electroacupuncture | Sham Electroacupuncture
Number analyzed (Participants) | 143 | 142
pmol/ml
  Change at week 8: number analyzed (Participants) | 143 | 141
  Change at week 8 | -12.3 [-59.5 to 35.0] | 19.5 [-38.5 to 77.6]
  Change at week 20: number analyzed (Participants) | 136 | 142
  Change at week 20 | -2.3 [-58.7 to 54.1] | -11.3 [-83.1 to 60.5]

14. Secondary Outcome: Change From Baseline in Serum LH Level
Description: The change from baseline in serum LH level at weeks 8 and 20 equals LH at weeks 8 and 20 minus LH at baseline, respectively.
Time Frame: at baseline, and weeks 8 and 20
Population: as for outcome 12
Measure: Mean (95% Confidence Interval); unit: mIU/ml
Arm/Group | Electroacupuncture | Sham Electroacupuncture
Number analyzed (Participants) | 171 | 172
mIU/ml
  Change at week 8 | 0.9 [-1.3 to 3.2] | 1.7 [-0.9 to 4.2]
  Change at week 20: number analyzed (Participants) | 164 | 166
  Change at week 20 | -1.3 [-4.2 to 1.6] | 0.1 [-2.6 to 2.8]

15. Secondary Outcome: Change From Baseline in Serum FSH/LH Level
Description: The change from baseline in serum FSH/LH at weeks 8 and 20 equals FSH/LH at weeks 8 and 20 minus FSH/LH at baseline, respectively.
Time Frame: at baseline, weeks 8 and 20
Population: as for outcome 12
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Electroacupuncture | Sham Electroacupuncture
Number analyzed (Participants) | 171 | 172
ratio
  Change at week 8 | 0.2 [0.1 to 0.3] | -0.1 [-0.3 to 0.0]
  Change at week 20: number analyzed (Participants) | 164 | 166
  Change at week 20 | 0.2 [0.0 to 0.3] | 0.0 [-0.1 to 0.1]

16. Secondary Outcome: Number of Participants Who Used Other Treatment During Study
Description: The number and percentage of patients who used other treatments will be compared between groups during weeks 1-8 and 9-32.
Time Frame: weeks 1-8; weeks 9-32
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Electroacupuncture | Sham Electroacupuncture
Number analyzed (Participants) | 174 | 175
Participants
  weeks 1- 8 | 8 | 8
  weeks 20-32: number analyzed (Participants) | 173 | 174
  weeks 20-32 | 7 | 9

ADVERSE EVENTS:
Time Frame: 32 weeks during the whole trial
Description: SAEs will be defined as events requiring hospitalization, causing disability or impaired ability to work, threatening life or resulting in death. AEs will be categorized as treatment related or non-treatment related based on its potential association with acupuncture needling procedure by acupuncturists and related specialists within 24 hours.
Groups:
- Sham Acupuncture: Electroacupuncture at non-points proximate to RN4 (P1), EX-CA1(P2)，ST25 (P3) and SP6 (P4) (double sides).One session will be given every two days, 3 sessions per week (24 sessions in all) and each session lasts for 30 minutes.sham acupuncture: Non-points proximate to RN4 (P1), EX-CA1(P2)，ST25 (P3) and SP6 (P4) (double sides) are used.P1 and P3 are at the sites 1 cm (outward in horizontal direction) proximate to RN4 and ST25 respectively. P2 is 2 cm (outward in horizontal direction) proximate to EX-CA1. P4 is at the middle site of the spleen meridian and the kidney meridian (backward in horizontal direction proximate to SP6).
  Stick adhesive tapes to all points. Blunt needles will be used to be inserted to but not piercing the skin. Even lifting, thrusting and twisting manipulation methods will be given for each non-point for 3 times. Put the sham electric stimulator on the pair of P2 and P3 with the same parameters as the acupuncture group. But there is no current intensity actually.
Arm/Group | Acupuncture | Sham Acupuncture
All-Cause Mortality (participants affected / at risk) | 0/180 | 0/180
Serious Adverse Events (participants affected / at risk) | 0/180 | 0/180
Other Adverse Events (participants affected / at risk) | 9/180 | 2/180
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acupuncture (N=180) | Sham Acupuncture (N=180)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Severe needling pain (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0)
Subcutaneous hematoma (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Fatigue (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Abdominal discomforts (Gastrointestinal disorders) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes